CLINICAL TRIAL: NCT02857205
Title: MICROPRUNG : Intestinal Microbiota Analysis in Patients With or Without Hirschsprung's Associated EnteroColitis
Acronym: MICROPRUNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC15_9873_MICROPRUNG; 2015-A01317-42 (Other: ANSM)
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung Associated EnteroColitis (HAEC)
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal samples (Other): High throughput sequencing methods and analysis for microbiome analysis on fecal samples from a multicenter cohort of patients at various ages.
  Interventions: Other: Fecal samples

INTERVENTIONS:
Other: Fecal samples — High throughput sequencing methods and analysis for microbiome analysis on fecal samples from a multicenter cohort of patients at various ages.

SUMMARY:
Hirschsprung disease is a congenital abnormality due to the lack of migration of neural crest cells in myenteric and submucosal plexi of the bowel wall. The consequence is the absence of parasympathetic control of the distal bowel from the anal sphincter to various levels. The most common type of Hirschsprung disease alters the rectosigmoid (80%). The incidence is around 1/5000 live births. This anomaly requires a surgical ablation of the aganglionic segment.

Regardless of the surgical complications, patients with Hirschsprung disease are exposed to the risk of Hirschsprung Associated EnteroColitis (HAEC). This variable risk, 4-54%, is responsible to a major part of Hirschsprung disease morbimortality. Its onset is more frequent during the first two years of life and then decrease with age.

Its pathogenesis remains unclear but could be due to intestinal homeostasis breakdown that involves microbiota, intestinal barrier, immune system and enteric nervous system. This breakdown of the mutual benefit relation due to microbiota or bowel anomaly is known to be responsible of Crohn's disease onset. Some studies emphasize the role of microbiota in the pathogenesis of HAEC, but the techniques or the methodology with small numbers of patients limit any conclusion or clinical use.

The study hypothesizes microbiota is a major factor in HAEC onset and in their functional bowel problems. Considering HAEC is more frequent the first two years, it's thought that intestinal microbiota changes with time in those patients. This project is innovative because it will use high throughput sequencing methods and analysis for microbiome analysis on fecal samples from a multicenter cohort of patients at various ages.

Multicentre transversal study.

This study has the potential to significantly modify clinical practice for Hirschsprung disease patients: a better care for HAEC and functional troubles thanks to a better understanding of their microbiota, targetted antibiotic treatment for HAEC, prophylactic treatment of patients at high risk of HAEC.

DETAILED DESCRIPTION:
Primary objective :

Characterize intestinal microbiota in patients with or without HAEC.

Secondary objectives :

* Look for a difference in microbiota composition between patients with or without HAEC ;
* Study the evolution with age of the microbiota in Hirschsprung disease patients ;
* Study predominant taxonomic classification elements in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 0 to 16 years ;
* With rectosigmoid Hirschsprung's disease confirmed by rectal biopsies and at surgery;
* Already operated on, whatever the surgical technique was ;
* With a health care insurance;
* Clear information and signed consent form

Exclusion Criteria:

* Long segment Hirschsprung disease ;
* Syndromic Hirschsprung disease ;
* Down syndrome.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiota composition | Sampling day
  Characterize intestinal microbiota in patients with or without HAEC

CONTACTS AND LOCATIONS:
Overall Officials: Alexis ARNAUD, MD, Principal Investigator — Rennes University Hospital
Locations (7):
- France (7):
  - Angers University Hospital, Angers
  - Brest University Hospital, Brest
  - Caen Univeristy Hospital, Caen
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No
Case Report Form

REFERENCES:
- [Derived] Arnaud AP, Cousin I, Schmitt F, Petit T, Parmentier B, Levard G, Podevin G, Guinot A, DeNapoli S, Hervieux E, Flaum V, De Vries P, Randuineau G, David-Le Gall S, Buffet-Bataillon S, Boudry G. Different Fecal Microbiota in Hirschsprung's Patients With and Without Associated Enterocolitis. Front Microbiol. 2022 Jun 30;13:904758. doi: 10.3389/fmicb.2022.904758. eCollection 2022. PMID 35847080